CLINICAL TRIAL: NCT02412371
Title: A Phase 1 Dose Escalation and Phase 2 Randomized, Placebo-Controlled Study of the Efficacy and Tolerability of Veliparib in Combination With Paclitaxel/Carboplatin-Based Chemoradiotherapy Followed by Veliparib and Paclitaxel/Carboplatin Consolidation in Subjects With Stage III Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study Evaluating the Efficacy and Tolerability of Veliparib in Combination With Paclitaxel/Carboplatin-Based Chemoradiotherapy Followed by Veliparib and Paclitaxel/Carboplatin Consolidation in Adults With Stage III Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase 2 was not conducted due to a change in the standard of care for newly diagnosed, unresectable Stage III NSCLC
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M14-360; 2016-001659-32 (EudraCT Number)
Record Dates: First submitted 2014-11-06; First posted 2015-04-09 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: veliparib; PARP inhibitor; ABT-888; first line; previously untreated; stage III; non-small cell lung cancer; radiotherapy; paclitaxel; carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; veliparib; Carboplatin; Radiotherapy

STUDY DESIGN:
Intervention Model Description: In the dose escalation phase (Phase 1) of the study participants will be enrolled sequentially to receive ascending dose of veliparib in combination with carboplatin + paclitaxel + thoracic radiotherapy.
  In the Phase 2 portion of the study participants were to be randomized in a 1:1:1 ratio to one of three treatment arms.
Masking Description: All participants will be treated with open-label paclitaxel and carboplatin (Phase 1 and Phase 2).
  Participants in Phase 1 will be treated with open-label veliparib. In Phase 2, the Sponsor, Investigator, study site personnel and participant were to be be blinded to each participant's treatment with veliparib or placebo throughout the course of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1: Veliparib + Carboplatin + Paclitaxel + Radiotherapy (Experimental): Participants in Phase 1 will be sequentially assigned to ascending dose levels of 60 mg, 80 mg, 120 mg, 200 mg, and 240 mg of twice daily (BID) veliparib in combination with carboplatin at an area under the concentration-time curve (AUC) 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent chemoradiotherapy participants will receive up to 2 cycles of consolidation therapy consisting of veliparib 120 mg or 240 mg BID, carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Veliparib; Radiation: Radiotherapy
- Phase 2: Veliparib + CRT -> Paclitaxel/Carboplatin/Veliparib (Experimental): Participants will receive veliparib at the recommended phase 2 dose determined in Phase 1 in combination with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent chemoradiotherapy participants will receive up to 2 cycles of consolidation therapy consisting of veliparib 120 mg or 240 mg BID, carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Veliparib; Radiation: Radiotherapy
- Phase 2: Veliparib + CRT -> Paclitaxel/Carboplatin/Placebo (Experimental): Participants will receive veliparib at the recommended phase 2 dose determined in Phase 1 in combination with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent chemoradiotherapy participants will receive up to 2 cycles of consolidation therapy consisting of placebo to veliparib BID, carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Paclitaxel; Drug: Placebo for Veliparib; Drug: Carboplatin; Drug: Veliparib; Radiation: Radiotherapy
- Phase 2: Placebo + CRT -> Paclitaxel/Carboplatin/Placebo (Active Comparator): Participants will receive placebo to veliparib with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent chemoradiotherapy participants will receive up to 2 cycles of consolidation therapy consisting of placebo to veliparib BID, carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Paclitaxel; Drug: Placebo for Veliparib; Drug: Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel — Administered via intravenous infusion on Day 1 of each treatment week (concurrent CRT) / cycle (consolidation)
Drug: Placebo for Veliparib — Capsule for oral administration
  Arms: Phase 2: Placebo + CRT -> Paclitaxel/Carboplatin/Placebo; Phase 2: Veliparib + CRT -> Paclitaxel/Carboplatin/Placebo
Drug: Carboplatin — Administered via intravenous infusion on Day 1 of each treatment week (concurrent CRT) / cycle (consolidation)
Drug: Veliparib — Capsule for oral administration
  Other Names: ABT-888
  Arms: Phase 1: Veliparib + Carboplatin + Paclitaxel + Radiotherapy; Phase 2: Veliparib + CRT -> Paclitaxel/Carboplatin/Placebo; Phase 2: Veliparib + CRT -> Paclitaxel/Carboplatin/Veliparib
Radiation: Radiotherapy — Radiation treatment with total dose of 60 - 63 Gy administered on Days 1 to 5 of each week for 7 weeks

SUMMARY:
This study seeks to establish

* the recommended Phase 2 dose (RPTD) of veliparib in combination with concurrent paclitaxel/carboplatin-based chemoradiotherapy (CRT) and consolidation with paclitaxel/carboplatin-based chemotherapy (Phase 1 portion), and
* to assess whether the addition of oral veliparib versus placebo to paclitaxel/carboplatin-based chemoradiotherapy with paclitaxel/carboplatin consolidation will improve progression-free survival (PFS) in adults with Stage III non-small cell lung cancer (Phase 2 portion).

A strategy decision was made not to proceed to Phase 2 portion of this study due to change in standard of care.

DETAILED DESCRIPTION:
This was to be a 2-phase study consisting of

1. A Phase 1, dose escalation study of veliparib to determine a RPTD for combination with concurrent paclitaxel/carboplatin-based CRT and paclitaxel/carboplatin-based consolidation chemotherapy; followed by
2. A Phase 2, randomized, double-blinded study to determine whether veliparib improved outcome relative to placebo when added to paclitaxel/carboplatin based CRT followed by consolidation paclitaxel/carboplatin in adults with previously untreated Stage III NSCLC.

In the dose escalation phase (Phase 1) of the study participants will be assigned to ascending doses of veliparib in combination with carboplatin, paclitaxel, and thoracic radiotherapy for 7 weeks following a traditional "3 + 3" design. The first cohort of at least 3 - 6 participants will receive veliparib 60 mg twice a day (BID) throughout CRT. Dose limiting toxicity (DLT) events will be collected for each dosing cohort until a new dosing cohort is opened or until the RPTD is identified. Participants will also receive a consolidation dose of veliparib of 120 mg BID + carboplatin and paclitaxel for up to two 21-day cycles. Once the concurrent CRT RPTD is identified, an additional cohort will be enrolled to explore the tolerability of a consolidation dose of veliparib at 240 mg BID + carboplatin + paclitaxel for up to two 21-day cycles.

Following the dose escalation portion of the study, the RPTD will be determined by the sponsor and the Phase 2 portion of the study will begin with patient randomization in a 1:1:1 ratio to concurrent paclitaxel/carboplatin/radiotherapy/veliparib followed by consolidation paclitaxel/carboplatin/veliparib, concurrent paclitaxel/carboplatin/radiotherapy/veliparib followed by consolidation paclitaxel/carboplatin/placebo, or concurrent paclitaxel/carboplatin/radiotherapy/placebo followed by consolidation paclitaxel/carboplatin/placebo. Randomization will be stratified by tumor volume (≤ 90 versus > 90 cm³) and smoking history (current smoker versus former smoker versus never smoked).

Phase 2 was not carried out since during the study there was a change in standard of care for patients with newly diagnosed, unresectable Stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with histologically or cytologically confirmed Stage III non-small cell lung cancer (NSCLC).
2. Participants in the randomized portion of the study must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 criteria.
3. Participants must have V20 (volume of lung to receive 20 Gy radiotherapy according to simulation) < 35%.
4. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance score of 0 - 1.
5. Participant must have adequate hematologic, renal, hepatic, and lung function.
6. Participant must consent to provide archived tissue or cytology sample of NSCLC lesion for analysis.

Exclusion Criteria:

1. Participants with prior chemotherapy or radiotherapy (RT) for current NSCLC. Participants curatively treated for past early stage NSCLC greater than 3 years ago may be included.
2. Participants with prior exposure to poly-adenosine diphosphate (ADP)-ribose polymerase (PARP) inhibitors.
3. Participants with known hypersensitivity to carboplatin, paclitaxel, or formulations containing polyethoxylated castor oil (Cremophor).
4. Participants with prior mediastinal or thoracic radiotherapy. Prior tangential radiotherapy to prior breast cancer is acceptable.
5. Participants with major surgery in the 4 weeks prior to randomization (Video-assisted thoracoscopic surgery (VATS) and/or mediastinoscopy is not considered major surgery).
6. Participants with a previous or concurrent malignancy except for treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient received potentially curative treatment and has been disease-free for 3 years or is considered cured by the investigator if has been disease-free for less than 3 years.
7. Participant is pregnant or lactating.
8. Participant with sensory peripheral neuropathy of ≥ Grade 2 at baseline, unable to swallow medication, or participants with prior history of seizure within the prior 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (12):
- United States (12):
  - Ucsd /Id# 133037, La Jolla, California
  - Christiana Care Health Service /ID# 133486, Newark, Delaware
  - University of Chicago /ID# 133828, Chicago, Illinois
  - Univ Maryland School Medicine /ID# 132944, Baltimore, Maryland
  - Dana-Farber Cancer Institute /ID# 133494, Boston, Massachusetts
  - SUNY Upstate Medical University - Downtown /ID# 133492, Syracuse, New York
  - Unc /Id# 133496, Chapel Hill, North Carolina
  - Duke University Medical Center /ID# 133497, Durham, North Carolina
  - Wake Forest Univ HS /ID# 134608, Winston-Salem, North Carolina
  - Rhode Island Hospital /ID# 133493, Providence, Rhode Island
  - The Miriam Hospital /ID# 133910, Providence, Rhode Island
  - University of Virginia /ID# 133495, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 48 participants at 10 sites in the United States. The study was designed as a 2-phase study consisting of a Phase 1, dose escalation of veliparib in combination with concurrent chemoradiotherapy (CRT) and consolidation chemotherapy (CT) and a Phase 2, randomized, double-blinded study.
Pre-assignment Details: Participants in Phase 1 were sequentially assigned to ascending dose levels of veliparib in combination with carboplatin/paclitaxel chemoradiotherapy. Phase 2 was not conducted since there was a change in standard of care for newly diagnosed, unresectable Stage III non-small cell lung cancer (NSCLC).
  Results are reported for Phase 1.
Groups:
- Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT: Participants received 60 mg veliparib twice daily (BID) in combination with carboplatin at an area under the concentration-time curve (AUC) 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy (RT) for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 120 mg BID with carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
- Veliparib 80 mg BID + CRT -> Veliparib 120 mg BID + CT: Participants received 80 mg veliparib BID in combination with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 120 mg BID with carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
- Veliparib 120 mg BID + CRT -> Veliparib 120 mg BID + CT: Participants received 120 mg veliparib BID in combination with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 120 mg BID with carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
- Veliparib 200 mg BID + CRT -> Veliparib 120 mg BID + CT: Participants received 200 mg veliparib BID in combination with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 120 mg BID, carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
- Veliparib 240 mg BID + CRT -> Veliparib 120 mg BID + CT: Participants received 240 mg veliparib BID in combination with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 120 mg BID with carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
- Veliparib 240 mg BID + CRT -> Veliparib 240 mg BID + CT: Participants received 240 mg veliparib BID in combination with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 240 mg BID, carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 80 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 120 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 200 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 240 mg BID + CT
Started | 7 | 9 | 7 | 8 | 12 | 5
Completed (Completed indicates participants remaining on study.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 9 | 7 | 8 | 12 | 5
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 1 | 0
Not completed — Sponsor Discontinued Study | 1 | 4 | 6 | 4 | 5 | 0
Not completed — Death | 4 | 2 | 1 | 3 | 5 | 2
Not completed — Other | 2 | 1 | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT: Participants received 60 mg veliparib BID in combination with carboplatin at an AUC 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 120 mg BID with carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 80 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 120 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 200 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 240 mg BID + CT | Total
Number analyzed (Participants) | 7 | 9 | 7 | 8 | 12 | 5 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (6.39) | 65.7 (7.55) | 66.9 (9.84) | 59.8 (6.07) | 67.3 (9.39) | 65.6 (11.84) | 65.8 (8.60)
Age, Customized [Count of Participants; unit: Participants]
  40 - < 60 years | 0 | 1 | 2 | 3 | 2 | 1 | 9
  ≥ 60 years | 7 | 8 | 5 | 5 | 10 | 4 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 5 | 6 | 5 | 3 | 29
  Male | 3 | 3 | 2 | 2 | 7 | 2 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 9 | 6 | 8 | 11 | 3 | 43
  Black | 1 | 0 | 1 | 0 | 1 | 2 | 5
Eastern Cooperative Oncology Group (ECOG) Performance Score [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis.
  * 0 = Fully Active (Most Favorable Activity);
  * 1 = Restricted activity but ambulatory;
  * 2 = Ambulatory but unable to carry out work activities;
  * 3 = Limited Self-Care;
  * 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    Grade 0 (Fully active) | 3 | 3 | 3 | 4 | 6 | 4 | 23
    Grade 1 (Restricted but ambulatory) | 4 | 6 | 4 | 4 | 6 | 1 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as the following events considered treatment-related by the Investigator, graded per Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
  * Radiation-induced myelopathy/myelitis or ≥ Grade (G) 3 cardiac toxicity
  * Radiation-related pneumonitis resulting in delay in RT, CT, or veliparib of >3 weeks or early discontinuation (DC) of RT (total dose <50 Gy)
  * ≥G4 esophagitis or esophagitis, dysphagia, and odynophagia requiring treatment interruption of >7 days despite medical management, neutropenia for >7 days or neutropenic fever or thrombocytopenia
  * ≥G2 seizure
  * G4 diarrhea or nausea/vomiting despite antiemetic therapy for >48 hours
  * Any other toxicity resulting in delay in RT, CT or veliparib >14 days or early DC of RT
  * Other nonhematologic toxicities ≥G3, except anorexia, fatigue, G3 infection, G3 aspartate/alanine transferase (AST/ALT) elevations ≤7 days, infusion reactions, G3/4 lymphopenia or electrolyte abnormalities corrected to ≤G2 in <48 hours
Time Frame: For Cohorts 1 - 5, from the start of veliparib dosing through 28 days after RT completion or until initiation of consolidation CT, approx. 10 weeks; For Cohort 6, 21 days from start of consolidation CT or until the start of cycle 2 consolidation therapy.
Population: Participants who received at least 1 dose of veliparib
Measure: Count of Participants; unit: Participants
Arm/Group | Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 80 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 120 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 200 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 240 mg BID + CT
Number analyzed (Participants) | 7 | 9 | 7 | 8 | 12 | 5
Participants | 0 | 0 | 0 | 1 | 0 | 2

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of participants who have a confirmed complete response (CR) or partial response (PR) as assessed by the investigator using RECIST v1.1. Participants who did not meet complete response or partial response, including those who did not have post-baseline radiological assessments were considered as non-responders.
  Complete Response (CR): The disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Normalization of tumor marker level. All lymph nodes must be non-pathological in size (< 10 mm short axis).
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Response must have been confirmed 4 weeks after the first documentation.
Time Frame: Tumor assessments were performed prior to consolidation chemotherapy, 24 weeks after start of treatment, every 8 weeks until 1 year after start of treatment, and then every 12 weeks until disease progression; median time on follow-up was 11 months.
Population: Participants who received at least 1 dose of veliparib and with at least one post-baseline tumor assessment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 80 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 120 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 200 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 240 mg BID + CT
Number analyzed (Participants) | 6 | 8 | 7 | 8 | 11 | 3
percentage of participants | 50.0 [11.8 to 88.2] | 50.0 [15.7 to 84.3] | 100.0 [59.0 to 100] | 62.5 [24.5 to 91.5] | 72.7 [39.0 to 94.0] | 0.0 [0.0 to 70.8]

3. Post Hoc Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from first dose of study drug to the date of earliest radiographic disease progression per investigator assessment based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death, and was calculated using Kaplan-Meier methods. All radiographic disease progression was included regardless whether the event occurred while the participant was taking study drug or had previously discontinued study drug. Participants who did not experience radiographic disease progression or death were censored at the date of the last disease assessment. Participants with no post-baseline disease assessment were censored at first dose date plus 1 day.
  Progressive disease (PD) was defined as at least a 20% increase in the size of target lesions with an absolute increase of at least 5 mm, unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
Time Frame: From first dose until end of study; maximum time on follow-up was approximately 46 months.
Population: All participants who received veliparib; PFS was pre-specified in the Protocol as a primary endpoint in Phase 2, which was not conducted. For Phase 1 PFS was not a pre-specified endpoint, and was only analyzed for all treatment cohorts combined due to the small sample sizes within each cohort.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Total: Participants received veliparib twice daily (BID) in combination with carboplatin at an area under the concentration-time curve (AUC) 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 120 or 240 mg BID with carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
Arm/Group | Total
Number analyzed (Participants) | 48
months | 19.6 [9.7 to 32.6]

4. Post Hoc Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from the participant's first dose of study drug to the date of death, and was calculated using Kaplan-Meier methods. Participants who did not die were censored at the date of last study visit or the last known date to be alive, whichever was later.
Time Frame: From first dose of study drug until end of study; maximum time on follow-up was approximately 46 months.
Population: All participants who received veliparib; OS was pre-specified in the Protocol as a secondary endpoint in Phase 2, which was not conducted. For Phase 1 OS was not a pre-specified endpoint, and was only analyzed for all treatment cohorts combined due to the small sample sizes within each cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Total
Number analyzed (Participants) | 48
months | 32.6 [15.0 to NA] — Could not be calculated due to the low number of events

5. Post Hoc Outcome: Duration of Overall Response (DOR)
Description: Duration of overall response was defined as time from the date of first response (CR or PR) to the earliest documentation of radiographic progressive disease or death due to disease progression, calculated using Kaplan-Meier methods. Participants who did not experience radiographic disease progression or death were censored at the date of the last disease assessment.
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of veliparib with at least 1 post-baseline tumor assessment and a confirmed response; DOR was prespecified as a secondary endpoint in Phase 2, which was not conducted. For Phase 1 DOR was not a prespecified endpoint and was only analyzed for all cohorts combined due to the small sample size of each cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Total
Number analyzed (Participants) | 27
months | 30.4 [17.5 to NA] — Could not be estimated due to the low number of events

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study drug to 30 days after the last dose of study drug; maximum duration of treatment was 14 weeks. Deaths were collected from the first dose of study drug through the end of study, up to 46 months.
Groups:
- Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT: Participants received 60 mg veliparib BID in combination with carboplatin at an area under the concentration-time curve (AUC) 2 mg/mL/min and paclitaxel 45 mg/m² once a week plus thoracic radiotherapy for 7 weeks.
  After completion of concurrent CRT participants received up to 2 cycles of consolidation therapy consisting of veliparib 120 mg BID with carboplatin AUC 6 mg/mL/min and paclitaxel 200 mg/m² administered on Day 1 of each 21-day cycle.
Arm/Group | Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 80 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 120 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 200 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 120 mg BID + CT | Veliparib 240 mg BID + CRT -> Veliparib 240 mg BID + CT
All-Cause Mortality (participants affected / at risk) | 5/7 | 3/9 | 1/7 | 3/8 | 6/12 | 3/5
Serious Adverse Events (participants affected / at risk) | 2/7 | 5/9 | 4/7 | 3/8 | 3/12 | 2/5
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9 | 7/7 | 8/8 | 12/12 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT (N=7) | Veliparib 80 mg BID + CRT -> Veliparib 120 mg BID + CT (N=9) | Veliparib 120 mg BID + CRT -> Veliparib 120 mg BID + CT (N=7) | Veliparib 200 mg BID + CRT -> Veliparib 120 mg BID + CT (N=8) | Veliparib 240 mg BID + CRT -> Veliparib 120 mg BID + CT (N=12) | Veliparib 240 mg BID + CRT -> Veliparib 240 mg BID + CT (N=5)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veliparib 60 mg BID + CRT -> Veliparib 120 mg BID + CT (N=7) | Veliparib 80 mg BID + CRT -> Veliparib 120 mg BID + CT (N=9) | Veliparib 120 mg BID + CRT -> Veliparib 120 mg BID + CT (N=7) | Veliparib 200 mg BID + CRT -> Veliparib 120 mg BID + CT (N=8) | Veliparib 240 mg BID + CRT -> Veliparib 120 mg BID + CT (N=12) | Veliparib 240 mg BID + CRT -> Veliparib 240 mg BID + CT (N=5)
ANAEMIA (Blood and lymphatic system disorders) | 3 (9) | 3 (4) | 3 (6) | 1 (3) | 6 (11) | 3 (10)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (3) | 4 (7) | 3 (12) | 2 (6) | 7 (16) | 4 (9)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (3) | 2 (5) | 1 (1) | 3 (4) | 5 (17) | 2 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (4) | 6 (7) | 6 (12) | 4 (6) | 9 (15) | 4 (7)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 6 (8) | 3 (7) | 3 (6) | 9 (18) | 4 (6)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EXTERNAL EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
VITREOUS FLOATERS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 4 (5) | 2 (2) | 2 (3) | 4 (9) | 3 (3) | 4 (5)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (4) | 1 (1) | 4 (6) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 5 (7) | 1 (1) | 4 (4) | 7 (12) | 3 (3) | 2 (3)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (4) | 5 (8) | 5 (10) | 4 (6) | 10 (16) | 5 (9)
ODYNOPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 4 (4) | 6 (7) | 4 (7) | 4 (5) | 9 (10) | 3 (4)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 4 (6) | 2 (3) | 2 (5) | 4 (7) | 3 (8)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CATHETER SITE PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
EXTRAVASATION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 6 (9) | 6 (6) | 5 (8) | 3 (3) | 7 (11) | 5 (7)
FEELING HOT (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GRAVITATIONAL OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE REACTION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOCALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MEDICAL DEVICE SITE ERYTHEMA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL DRYNESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERFORMANCE STATUS DECREASED (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 1 (1)
SWELLING FACE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATHETER SITE CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX OESOPHAGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RADIATION INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RADIATION OESOPHAGITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 2 (2) | 2 (3) | 3 (4) | 3 (5) | 5 (11) | 4 (5)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 3 (3) | 2 (2) | 2 (6) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (5) | 2 (3) | 5 (5) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 1 (5) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (3) | 2 (3) | 4 (6) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 4 (4) | 1 (1)
DIZZINESS POSTURAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (3) | 3 (6) | 4 (4) | 1 (2) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (4) | 1 (1) | 2 (3) | 2 (3) | 1 (1) | 2 (4)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TASTE DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
NERVOUSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL RASH (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 3 (4) | 2 (2)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT02412371/Prot_SAP_000.pdf